CLINICAL TRIAL: NCT04078191
Title: A Comparison of Tc 99m Tilmanocept Quantitative Imaging With Immunohistochemical (IHC) Analysis of CD206 Expression in Synovial Tissue From Subjects Clinically Diagnosed With Rheumatoid Arthritis (RA)
Brief Title: Comparison of Tc 99m Tilmanocept Imaging With IHC Analysis of CD206 Expression in Synovial Tissue of Subjects With RA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-32; 2018-003418-41 (EudraCT Number)
Record Dates: First submitted 2019-08-21; First posted 2019-09-04 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
Keywords: tilmanocept; RA imaging; synovial biopsy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RA Subjects on Stable Therapy (Experimental): RA subjects who are on stable treatment will receive a single dose of 150 mcg tilmanocept radiolabeled with 10 mCi Tc 99m.
  Interventions: Drug: Tc 99m tilmanocept

INTERVENTIONS:
Drug: Tc 99m tilmanocept — Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Other Names: Lymphoseek

SUMMARY:
This study is a comparison of quantitative Tc 99m tilmanocept imaging with IHC analysis of CD206 expression in synovial tissue of RA subjects.

DETAILED DESCRIPTION:
This is a Manocept Platform phase 2b, open-label, multi-center, multinational, non-randomized, single-dose study designed to assess the relationship between quantitative Tc 99m tilmanocept planar imaging and synovial histopathology in subjects clinically diagnosed with RA.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has provided written informed consent with HIPAA (Health Information Portability and Accountability Act) or equivalent authorization before the initiation of any study-related procedures.
2. Women and men of childbearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) for the duration of the study.
3. The subject is at least 18 years of age and was ≥ 18 years of age at the time of RA diagnosis.
4. The subject has RA as determined by the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Classification Criteria (score of ≥ 6/10 at or before screening).
5. The subject has a 28-joint disease activity score (DAS28) of ≥ 3.2 (includes the C-reactive protein [CRP] test and visual analog scale [VAS]).
6. Subjects receiving traditional DMARDs must have been on therapy for ≥ 90 days and at a stable dose for ≥ 30 days prior to the first imaging visit (Day 0).
7. If the subject is receiving biologic disease-modifying antirheumatic drug (bDMARD) or janus kinase (JAK) inhibitor therapy, they have been at a stable dose > 180 days prior to the first imaging visit (Day 0).
8. If the subject is receiving NSAIDs (nonsteroidal anti-inflammatory drug) or oral corticosteroids, the dose has been at a stable dose for ≥ 28 days prior to imaging. The corticosteroid dose should be ≤ 10 mg/day of prednisone or an equivalent steroid dose.
9. The subject has a hand or wrist joint with a minimum ultrasound gray-scale synovitis score of 2 (range 0 to 3).

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject size or weight is not compatible with imaging per the investigator.
3. The subject has had or is currently receiving radiation therapy or chemotherapy.
4. The subject has renal insufficiency as demonstrated by a glomerular filtration rate of < 60 mL/min.
5. The subject has hepatic insufficiency as demonstrated by ALT (alanine aminotransferase [SGPT]) or AST (aspartate aminotransferase [SGOT]) greater than 3 times the upper limit of normal.
6. The subject has any severe, acute, or chronic medical conditions and/or psychiatric conditions and/or laboratory abnormalities that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration that would deem the subject inappropriate for study participation.
7. The subject has a known allergy to or has had an adverse reaction to dextran exposure.
8. The subject has received an investigational product within 30 days prior to the Tc 99m tilmanocept administration (Day 0).
9. The subject has received intra-articular corticosteroids ≤ 8 weeks prior to imaging (Day 0).
10. The subject has received any radiopharmaceutical within 7 days or 10 half-lives prior to the administration of Tc 99m tilmanocept (Day 0).
11. The subject has an intolerance to anesthetic and antiseptic agents indicated for the synovial biopsy procedure.
12. The subject is currently receiving anticoagulants (oral anti-platelet agents are permitted) or has a condition that is contraindicated with ultrasound-guided synovial biopsy e.g., needle phobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Study Director — Navidea Biopharmaceuticals
Locations (4):
- United States (2):
  - Attune Health, Beverly Hills, California
  - Northwestern University, Chicago, Illinois
- United Kingdom (2):
  - Barts Hospital, London, England
  - Royal Free Hospital, London, England

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RA Subjects on Stable Therapy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RA Subjects on Stable Therapy
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 59.0 [24 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13
  United Kingdom | 7

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Joint-specific Tilmanocept Uptake and CD206 Expression
Description: The correlation between joint-specific tilmanocept uptake value (TUVjoint) and the number and area fraction of CD206 expression as determined by IHC assessment.
Time Frame: Through study completion, up to 45 days
Population: Data not collected.
Arm/Group | RA Subjects on Stable Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Correlation Between Joint-specific Tilmanocept Uptake and CD68 and CD163 Expression
Description: The correlation between TUVjoint and the number and area fraction of CD68 and CD163 determined by IHC assessments.
Time Frame: Through study completion, up to 45 days
Population: Data not collected.
Arm/Group | RA Subjects on Stable Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Classification of Synovial Anatomic Pathotype by IHC Assessment
Description: Classification of synovial anatomic pathology into
  * Lympho-myeloid
  * Diffuse myeloid
  * Pauci-immune fibroid types as a function of CD68, CD163, CD206, CD3, CD20, CD55, and TE7 expression determined by IHC assessments using a polytomous logistic regression model.
Time Frame: Through study completion, up to 45 days
Population: All enrolled subjects injected with Tc99m technetium
Measure: Count of Participants; unit: Participants
Arm/Group | RA Subjects on Stable Therapy
Number analyzed (Participants) | 20
Participants
  Pauci-immune/Fibroid | 8
  Diffuse/Myeloid | 8
  Lympho-Myeloid | 4

4. Other Pre Specified Outcome: Exploratory Objective: Correlation Between CD206, CD68, and CD163 Expression
Description: * Determine the relationship between TUVjoint and mRNA expression profiles of CD68, CD163, and CD206 as determined by RNA sequencing (RNA-seq).
  * Determine the relationship between TUVjoint and the number, size, and intensity of CD68, CD163, and CD206 as determined by (optional) flow cytometry.
  * Evaluate synovial expression of CD3, CD20, CD55, and TE-7 and CD206 in synovial tissue biopsy specimens.
  * Assessment of the relationship between TUVglobal and synovial anatomic pathology.
Time Frame: Through study completion, up to 45 days
Population: Data not collected.
Arm/Group | RA Subjects on Stable Therapy
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Safety Evaluation - AEs
Description: Evaluate safety through the examination of adverse event (AE) incidence.
Time Frame: Through study completion, up to 45 days
Population: All enrolled subjects injected with Tc99m technetium.
Measure: Number; unit: Adverse Events
Arm/Group | RA Subjects on Stable Therapy
Number analyzed (Participants) | 20
Adverse Events
  Adverse Events | 25
  Serious Adverse Events | 1

6. Other Pre Specified Outcome: Safety Evaluation - Laboratory Tests, ECGs, and Vital Signs
Description: Evaluate safety through physical examination findings, and changes over time in laboratory tests, electrocardiograms (ECGs), and vital signs.
Time Frame: Through study completion, up to 45 days
Population: All enrolled subjects injected with Tc99m technetium.
Measure: Number; unit: Incidents
Arm/Group | RA Subjects on Stable Therapy
Number analyzed (Participants) | 20
Incidents
  Clinically Significant Laboratory Tests | 0
  Clinically Significant ECG Readings | 0
  Clinically Significant Vital Signs | 0

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | RA Subjects on Stable Therapy
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA Subjects on Stable Therapy (N=20)
Covid (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Covid Infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA Subjects on Stable Therapy (N=20)
Pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Fever (Immune system disorders) | 1 (1)
Swelling (Musculoskeletal and connective tissue disorders) | 6 (6)
Bruising (Musculoskeletal and connective tissue disorders) | 5 (14)
Headache (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Trouble falling asleep (Psychiatric disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Analysis of NAV3-32 trial data was halted prior to evaluation of the acquired images. Preliminary analysis of data from other trials indicated that the ability of Tc 99m tilmanocept imaging to predict response to anti-TNFα therapy in RA patients would not be sufficient for the product to be commercially viable. Therefore, further development of the product for this indication was halted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trail Agreement prevents any PIs to publish data that has not been approved by the sponsor.

DOCUMENTS (3):
  • Study Protocol (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT04078191/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT04078191/SAP_002.pdf
  • Informed Consent Form (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT04078191/ICF_001.pdf